CLINICAL TRIAL: NCT03373890
Title: Muscle Performance and Walking in Cerebral Palsy: Short-burst Interval Training
Brief Title: Cerebral Palsy: Short-burst Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Kristie Bjornson, Associate Professor, Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD077186 (NIH)
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Palsy Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Pre/post intervention design with participants randomized to two different frequency of intervention
Who Masked: Outcomes Assessor
Masking Description: Muscle function assessor masked to frequency group, Muscle architecture captured via ultrasound Community walking activity collected by accelerometry, thus non-human data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short burst Interval Treadmill Training High Frequency (Experimental): Participants receive short burst interval treadmill training for a total of 20 sessions. They are randomized to receive it either 5x/week for 4 weeks
  Interventions: Behavioral: Short Burst Interval Locomotor Treadmill Training (SBLTT)
- Short Burst Interval Treadmill Training Low Frequency (Active Comparator): Participants receive short burst interval treadmill training for a total of 20 sessions. They are randomized to receive it either 2x/week for 10 weeks
  Interventions: Behavioral: Short Burst Interval Locomotor Treadmill Training (SBLTT)

INTERVENTIONS:
Behavioral: Short Burst Interval Locomotor Treadmill Training (SBLTT) — SBLTT consists of interval training consisting of short-bursts (30 seconds) of vigorous intensity locomotor treadmill training (LTT) alternating with low to moderate intensity LTT.,

SUMMARY:
This study examines the effect of short burst interval treadmill training in ambulatory children with cerebral palsy. Half the sample will receive 20 sessions of training over 4 weeks, while half will receive the training over 10 weeks.

DETAILED DESCRIPTION:
Ambulatory children with cerebral palsy (CP) experience activity limitations which negatively influence their ability to physically participate in day to day life. Therefore, these children are at greater risk for inactivity and functional decline with age. In contrast, typically developing (TD) children engage in short bursts of intense physical activity interspersed with varying intervals of low and moderate intensity within their natural environment. These physical activity patterns are very different from adult patterns Despite these inherent differences, locomotor treadmill training (LTT) protocols designed to improve walking activity in children with CP simulate adult protocols, consisting of continuous low to moderate walking endurance activity. Body weight supported or robot assisted LTT is based on the underlying premise of modifying neural circuitry via spinal pathways. However, this type of training has not been shown to be more effective than other comparable interventions and presents with significant fiscal and logistical barriers to clinical translation.

This study will determine the effect of short-burst interval LTT without body weight support on the primary outcomes of walking performance and capacity and the secondary outcomes of day-to-day mobility based participation in children with CP with functional walking limitations. To identify key muscular mechanisms associated with improved walking mobility, the investigators will examine the effects of short-burst interval LTT on quadriceps muscle performance and architecture. Secondarily, the study team will collect preliminary data on two LTT dosing frequencies.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory children with cerebral palsy Spasticity primary movement disorder Bilateral motor impairment (Diplegia) Gross Motor Function Classification System Levels II and III

Exclusion Criteria:

* undergone orthopedic or neurosurgery less than 12 months prior injection therapies (phenol, botulinum toxin) less than 3 months prior

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Hendricks, PhD, Study Director — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a directed mailing to children with cerebral palsy receiving care at Seattle Children's Hospital between Sept 1, 2014 and June 30 2015.
Pre-assignment Details: In eligible if unable to walk at greater than their self selected walking speeds with orthotics on a treadmill.
Groups:
- Short Burst Interval Treadmill Training High Frequency: All participants receive short burst interval treadmill training for a total of 20 sessions. They are randomized to receive 5x/week for 4 weeks.
  Short Burst Interval Locomotor Treadmill Training (SBLTT): SBLTT consists of interval training consisting of short-bursts (30 seconds) of vigorous intensity locomotor treadmill training (LTT) alternating with low to moderate intensity LTT.
- Short Burst Interval Treadmill Training Low Frequency: All participants receive short burst interval treadmill training for a total of 20 sessions. They are randomized to receive 2 x/week for10 weeks.
  Short Burst Interval Locomotor Treadmill Training (SBLTT): SBLTT consists of interval training consisting of short-bursts (30 seconds) of vigorous intensity locomotor treadmill training (LTT) alternating with low to moderate intensity LTT.
Period: Overall Study
Arm/Group | Short Burst Interval Treadmill Training High Frequency | Short Burst Interval Treadmill Training Low Frequency
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Short Burst Interval Treadmill Training High Frequency: All participants receive short burst interval treadmill training for a total of 20 sessions. They are randomized to receive it either 5x/week for 4 weeks
  Short Burst Interval Locomotor Treadmill Training (SBLTT): SBLTT consists of interval training consisting of short-bursts (30 seconds) of vigorous intensity locomotor treadmill training (LTT) alternating with low to moderate intensity LTT.
- Short Burst Interval Treadmill Training Low Frequency: All participants receive short burst interval treadmill training for a total of 20 sessions. They are randomized to receive it either 2x/week for 10 weeks
  Short Burst Interval Locomotor Treadmill Training (SBLTT): SBLTT consists of interval training consisting of short-bursts (30 seconds) of vigorous intensity locomotor treadmill training (LTT) alternating with low to moderate intensity LTT.
- Total: Total of all reporting groups
Arm/Group | Short Burst Interval Treadmill Training High Frequency | Short Burst Interval Treadmill Training Low Frequency | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (2.3) | 9.4 (2.0) | 8.6 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All participants lived in western Washington state.
  participants
    United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Performance High Versus Low Frequency SBLTT Groups
Description: Average stride per day as measured by StepWatch accelerometry. StepWatch accelerometer stride counts per day ( minimum of 8 hrs/day wearing time) were averaged a crossed 5 days (4 weekdays and 1 weekend day) to create Average Strides/day variable
Time Frame: Change from baseline to immediately post SBLTT
Population: Change in average strides/day from baseline to immediately post SBLTT were compared between the high and low frequency groups/arms.
Measure: Mean (Standard Deviation); unit: strides per day
Groups:
- High Frequency 5x/Week: This group received short burst interval treadmill training 5x/week for total of 20 sessions
- Low Frequency 2x Week: Received short burst interval training 2x week for total of 20 sessions
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
strides per day | 1872 (880) | 1551 (952)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — Independent samples Mann Whitney U; p = .39, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Community Walking Performance Intensity High Versus Low Frequency SBLTT Groups
Description: Average Strides/day > 30 strides/min as measured by StepWatch accelerometry High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to immediately post SBLTT
Population: Change in average strides/day > 30 strides/min as measured by StepWatch accelerometry for one side a cross 5 days (4 weekdays and 1 weekend day)
Measure: Mean (Standard Error); unit: strides per day
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
strides per day | 866 (652) | 731 (522)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — Independent samples Mann Whitney U; p = .39, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Walking Capacity High Versus Low Frequency SBLTT Groups
Description: Self selected walking speed as measured by 10 meter walk test High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to immediately post SBLT.
Population: Change in self selected walking speed between baseline and immediately post SBLTT was compared between the high and low frequency groups/arms.
Measure: Mean (Standard Deviation); unit: meters per sec
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
meters per sec | .21 (.3) | -.08 (.2)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — Independent samples Mann Whitney U; p = .03, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Walking Endurance- High Versus Low Frequency SBLTT Groups
Description: Distance walked during the One Minute Walk Test High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to immediately post SBLTT
Population: Change in distance walked in one minute between baseline and immediately post SBLTT compared between high and low frequency groups.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
meters | 13.8 (2.5) | 8.8 (2.6)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — Independent samples Mann Whitney U; p = .39, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Muscle Performance -Power High Versus Low Frequency SBLTT Groups
Description: Knee extensor muscle power - isotonic muscle power as measured by Biodex testing High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to 6 weeks post SBLTT
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
watts | 1.2 (.11) | 1.9 (.19)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — Independent samples Mann Whitney U; p = .06, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Muscle Performance - Strength High Versus Low Frequency SBLTT Groups
Description: Knee extensor muscle strength - isometric muscle strength as measured by Biodex testing High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to immediately post SBLTT
Population: Change in normalized isometric quadriceps strength as measured by Biodex, from baseline to immediately post SBLTT compared between high and low frequency groups/arms.
Measure: Mean (Standard Deviation); unit: newton meters
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
newton meters | .13 (.25) | .14 (.50)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — Independent samples Mann Whitney U; p = .99, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Muscle Architecture-High Versus Low Frequency SBLTT Groups
Description: Rectus femoris mid thigh cross-sectional area as measured by 2D B Mode Ultrasound High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to immediately post SBLTT
Population: Change in rectus femoris cross sectional area as measured by 2D B Mode ultrasound, from baseline to immediately post SBLTT compared between high and low frequency groups/arms.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
Number analyzed (Participants) | 6 | 6
mm^2 | .05 (.02) | 0 (.03)
Statistical Analysis 1: Comparison: High Frequency 5x/Week vs Low Frequency 2x Week; Test type: Other — LInear mixed model; p = .008, Regression, Logistic

8. Secondary Outcome: Change in Muscle Architecture-hypertrophy High Versus Low Frequency SBLTT Groups
Description: Rectus femoris mid thigh fascicle length as measured by 2D B Mode Ultrasound High Versus Low Frequency SBLTT Groups
Time Frame: Change from baseline to immediately post SBLTT
Population: Change in rectus femoris mid thigh fascicle length as measured by 2D B Mode ultrasound , from baseline to immediately post SBLTT compared between high and low frequency groups/arms.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Short Burst Interval Treadmill Training High Frequency | Short Burst Interval Treadmill Training Low Frequency
Number analyzed (Participants) | 6 | 6
millimeters | .06 (.12) | .05 (.13)
Statistical Analysis 1: Comparison: Short Burst Interval Treadmill Training High Frequency vs Short Burst Interval Treadmill Training Low Frequency; Test type: Other — Linear mixed model regression; p = .34, Regression, Linear

ADVERSE EVENTS:
Time Frame: Reported from consent/baseline to 6 week post intervention follow up which for high frequency group was approximately 4 months and for the low frequency group was 6 months
Description: Severity coded Mild, moderate or severe Mild= inconvenience to day to day life Moderate= required medical attention Severe= Life threatening
  Relationship to study:
  Definitely Not Possibly Definitely Related
Arm/Group | High Frequency 5x/Week | Low Frequency 2x Week
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Frequency 5x/Week (N=6) | Low Frequency 2x Week (N=6)
Mild severity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — fall while walking down stairs at home not during treadmill training
Mild possibly related to study (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — blister from new Ankle Foot Orthoses (AFO)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No